CLINICAL TRIAL: NCT07089953
Title: Patient Perception of Physician's Compassion, Communication Skills, and Professionalism During Clinic Visits: a Randomized Controlled Trial (EHR Study #3)
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0651; NCI-2025-05414 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Communication Skills; Professionalism; Randomized Controlled Trial; Perception
MeSH Terms: interventions — Surveys and Questionnaires; Videotape Recording

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1: Physician A - No EHR
  Interventions: Other: Questionnaire; Other: Video
- Arm 2: Physician B - No EHR
  Interventions: Other: Questionnaire; Other: Video
- Arm 3: Physician A - Prime EHR
  Interventions: Other: Questionnaire; Other: Video
- Arm 4: Physician B - Prime EHR
  Interventions: Other: Questionnaire; Other: Video

INTERVENTIONS:
Other: Questionnaire — Complete 3 questionnaires about your emotions and your trust in doctors.
  Other Names: Questionnaires/Survey Measures
Other: Video — Four (4) videos, each 4 minutes long, have been made for use in this study.

SUMMARY:
To learn about how patients view a doctor's compassion, communication skills, and professionalism based on whether the doctor uses the Electronic Health Record (EHR) during a visit with a patient.

DETAILED DESCRIPTION:
Primary Objectives 1. To compare participants' perception of physicians' compassion after they watch two scripted-video vignettes of physicians: one portraying a traditional face to face clinical visit without the use of examination room computer, and the other one portraying a physician using an integrated model of EHR use for communication during the visit.

Secondary Objectives

1. Study To compare participants' perception of physicians' communication skills after they watch two scripted-video vignettes of physicians: one portraying a traditional face to face clinical visit without examination room computer use, and the other one portraying a physician using an integrated model of EHR use during communication.

ELIGIBILITY:
Eligibility Criteria

1. Participants with a diagnosis of cancer either early disease or advanced cancer defined as locally advanced, recurrent, or metastatic disease.
2. Outparticipants (either new referrals or follow-ups) seen in the Supportive Care Clinic.
3. Age >/= 18 years old.
4. Able to read, write, and speak English.
5. Participants with normal cognitive status (Memorial Delirium Assessment Scale (MDAS) </= 6/30) who can understand the nature and purpose of the study and have the ability to complete the consent process.

Exclusion Criteria

1. Participants who are experiencing severe symptom distress, including severe emotional distress, which may interfere with study participation. This will be measured by the Edmonton Symptom Assessment Scale (ESAS). Eligibility of participants with ESAS score >/= 7 on any item will be determined by the principal investigator and/or attending physician who is caring for the patient during that visit.
2. Participants with cognitive dysfunction (Memorial Delirium Assessment Scale (MDAS) >/= 7/30 will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaires/Videos | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ali Haider, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States